CLINICAL TRIAL: NCT06325761
Title: A Randomized, Open-label, Single-dose, Two-period, Two-treatment Crossover Study Evaluating the Effects of Food on the Pharmacokinetics of SY-5007 Tablets in Chinese Healthy Subjects
Brief Title: A Study to Evaluate the Food Effects on Pharmacokinetics of SY-5007 Tablets in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shouyao Holdings (Beijing) Co. LTD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SY-5007-I-02
Record Dates: First submitted 2024-03-13; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Health Subjects
Keywords: SY-5007 tablets; Food effect; Two-period crossover

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasted dosing followed by fed dosing (Experimental): A single oral dose in the fasted state at Period 1 followed by fed dosing at Period 2
  Interventions: Drug: SY-5007
- Fed dosing followed by fasted dosing (Experimental): A single oral dose in the fed state at Period 1 followed by fasted dosing at Period 2
  Interventions: Drug: SY-5007

INTERVENTIONS:
Drug: SY-5007 — SY-5007 160 mg, Tablets, 2 discrete single doses separated by 7-days
  Arms: Fasted dosing followed by fed dosing
Drug: SY-5007 — SY-5007 160 mg, Tablets, 2 discrete single doses separated by 7-days
  Arms: Fed dosing followed by fasted dosing

SUMMARY:
This study is a single-center, randomized, open-label, single-dose, two-period, two-treatment crossover trial aimed at evaluating the pharmacokinetic (PK) profiles and safety of SY-5007 tablets administered orally to healthy subjects in both fasting and fed states in China.

DETAILED DESCRIPTION:
The study consists of two parts: a pilot study and a formal study. The pilot study involves four healthy subjects who will receive a single dose of SY-5007 80 mg after a meal (high-fat meal) for Period 1 and on an empty stomach for Period 2, with observation and PK blood sample collection.

The formal study plans to enroll 24 healthy subjects, divided into Groups A and B, each with 12 subjects, receiving a dose of 160 mg. Group A will receive the drug on an empty stomach for Period 1, followed by administration after a meal (high-fat meal) for Period 2, while Group B will follow the reverse sequence. Both groups will adopt a two-period, two-treatment crossover design with a washout period of 7 days. If the pilot study results show a significant impact of food on the PK characteristics or safety of SY-5007, subsequent trial protocols may be adjusted.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for participation in this study:

1. Fully understand the purpose, nature, methods, and potential adverse reactions of the trial, voluntarily participate, and sign a written informed consent form (ICF), and be able to follow the protocol requirements to complete the study as healthy subjects.
2. Aged ≥18 and ≤55 years old, regardless of gender (including boundary values, based on the time of signing the informed consent form).
3. Male subjects with a body weight ≥50kg, female subjects with a body weight ≥45kg, and a body mass index (BMI = weight/height^2, kg/m^2) between 18 and 26 kg/m^2 (including boundary values).
4. Female subjects of childbearing potential and all male subjects agree to adopt effective contraception with their sexual partners during the study and for 3 months after the last dose, and have no plans to donate sperm/eggs during the trial and for 3 months after the end of the trial.

Exclusion Criteria:

Subjects will be ineligible for this study if they meet any of the following criteria:

1. A clear history of severe allergies, non-allergic drug reactions, or multiple drug allergies, or known hypersensitivity reactions to the investigational drug (active pharmaceutical ingredient or excipients).
2. Positive for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen, hepatitis C antibodies, or syphilis treponema antibodies at screening.
3. Clinically significant abnormal vital signs, physical examination findings, laboratory test results, or electrocardiogram results at screening.
4. Currently suffering from or known by the investigator to have chronic gastrointestinal, liver, or kidney diseases that may affect trial outcomes.
5. Any symptoms or medical history of major diseases within the past two years, including but not limited to cardiovascular, hepatic, renal diseases, or other acute or chronic gastrointestinal diseases, respiratory diseases, musculoskeletal diseases, as well as diseases of the blood, endocrine, nervous, or psychiatric systems, or any other conditions or physiological states that may interfere with trial results.
6. Any surgical conditions or conditions that may significantly affect drug absorption, distribution, metabolism, and excretion, or any surgical conditions or conditions that may pose harm to subjects participating in the trial, such as a history of gastrointestinal surgery (gastrectomy, gastrojejunal anastomosis, intestinal resection, etc.), urinary tract obstruction or difficulty in urination, history of digestive tract ulcers, gastrointestinal bleeding, etc. (Subjects who have undergone appendectomy or hernia repair surgery can be enrolled in the study).
7. Known or suspected history of drug abuse within the past two years at screening, or drug abuse within the past three months at screening or baseline, or positive drug abuse screening during screening or baseline.
8. Underwent major surgery within the past six months before the first dose or planning to undergo surgery during the trial.
9. Smoked an average of more than 5 cigarettes per day within the past three months before the first dose or unwilling to stop using any tobacco products during the trial.
10. Regularly consumed alcohol within the past three months before the first dose (defined as consuming more than 14 units of alcohol per week, with 1 unit equal to 360 mL of beer with an alcohol content of 5%, or 45 mL of spirits with an alcohol content of 40%, or 150 mL of wine with an alcohol content of 12%), or unable to stop drinking during the trial, or positive alcohol breath test at screening.
11. History of blood donation or significant blood loss (≥300 mL) within the past two years before the first dose, or use of blood products or receiving blood transfusions within the past month before the first dose.
12. Participated in other drug or medical device clinical trials within the past three months before the first dose (excluding those screened but ultimately not enrolled), or used the study drug before.
13. Received vaccination or inactivated vaccines within the past month before the first dose.
14. Used any prescription drugs, non-prescription drugs, health products, or herbal medicines within the past two weeks before the first dose (if the half-life (t1/2) of the drug used can be confirmed, the washout period should be ≥5 t1/2, with the longer one taken).
15. Habitually consumed grapefruit juice or excessive amounts (more than 8 cups, 1 cup = 250 mL) of tea, coffee, and/or caffeinated beverages and unable to stop drinking for at least 48 hours before the first dose and during the trial.
16. Have special dietary requirements or difficulty swallowing.
17. Difficulty in blood sampling, or a history of fainting or intolerance to venipuncture.
18. A clear history of neurological or psychiatric disorders, including dementia or epilepsy, etc.
19. Diagnosis of malignant tumors within the past five years (excluding cured in situ cancers, such as non-melanoma skin cancers).
20. For scientific reasons, compliance reasons, or for the safety of the subjects, the investigator deems it inappropriate for the subject to participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Cmax for SY-5007 | Day 1-Day 15
  Defined as maximum observed plasma concentration
Tmax for SY-5007 | Day 1-Day 15
  Defined as time to maximum plasma concentration
AUC0-t for SY-5007 | Day 1-Day 15
  Defined as area under the single-dose plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration
AUC0-∞ for SY-5007 | Day 1-Day 15
  Defined as area under the single-dose plasma concentration-time curve from Hour 0 to infinity
t½ for SY-5007 | Day 1-Day 15
  Defined as apparent plasma terminal phase disposition half-life
CL/F for SY-5007 | Day 1-Day 15
  Defined as apparent total body clearance
Vz/F for SY-5007 | Day 1-Day 15
  Defined as apparent oral Volume of distribution

SECONDARY OUTCOMES:
Safety of SY-5007 | Day 1-Day 22
  AE (adverse event) will be summarized by type and severity

CONTACTS AND LOCATIONS:
Overall Officials: Yinghui Sun, Dr, Study Director — Shouyao Holdings (Beijing) Co. LTD
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China